CLINICAL TRIAL: NCT05959902
Title: Effectiveness of Physical Therapy on Stem Cell Transplantation Recipients in Improving Pain, Quadriceps Muscle Strength and Functional Status of Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: Effectiveness of Physical Therapy in Stem Cell Transplant Recipients for Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Syed Muhammad Zaeem Hasan Zaidi, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2777
Record Dates: First submitted 2023-07-16; First posted 2023-07-25 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis; Osteo Arthritis Knee; OA Knee
Keywords: Knee osteoarthritis; Mesenchymal stem cell treatment; Physiotherapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forward Walking (Active Comparator): This study ARM will receive following treatment in home program after mesenchymal stem cell treatment.
  • Forward Walking
  Interventions: Other: Forward Walking
- Physiotherapy (Experimental): This study ARM will be receiving following physiotherapy exercises for knee osteoarthritis after mesenchymal stem cell therapy.
  * Isometric quadriceps exercise
  * Straight leg raising (SLR) exercise
  * Isometric hip adduction exercise
  * Terminal knee extension exercise
  * Semi wall squat exercise
  * Quadriceps drill exercise
  Interventions: Other: Physiotherapy Exercises

INTERVENTIONS:
Other: Forward Walking — During the 8-week treatment, the participants will undertake 10 minutes of forward walking, as well as a 5-minute warm-up and cool-down, three times a week on an even surface at their normal speed as a home exercise plan. During the warmup and cool down periods, the participants were advised to execute ankle toe motions, heel lift exercises, and hamstring and gastrocnemius-soleus stretches.
  Arms: Forward Walking
Other: Physiotherapy Exercises — Isometric quadriceps exercise. Straight leg raising (SLR) exercise. Isometric hip adduction exercise.
  Terminal knee extension exercise:
  Semi-wall squat exercise. Quadriceps drill exercise.
  Arms: Physiotherapy

SUMMARY:
Knee osteoarthritis has been considered as 11th highest contributor factor to nonfatal burdens in the world. It is considered one of the most common degenerative diseases of synovial joint and major cause of muscle impairment with limited functional activities. Recent efforts to investigate the possibility of stem cell therapies in the treatment of symptomatic osteoarthritis have seen an increase in interest in regenerative medicine, fueled a better understanding of the role of mesenchymal stem cells. Knee osteoarthritis is mostly managed by physical therapy, focused on managing pain, increasing the restricted range of motion and muscle strengthening. Therefore, the hypothesis is that combining both treatments will be beneficial for patients. The aim of this randomized controlled trial is to evaluate the effectiveness of physiotherapy in mesenchymal stem cell recipient in improving pain, quadriceps muscle strength and functional status of knee osteoarthritis patients.

DETAILED DESCRIPTION:
A single blinded RCT will be conducted at Ortho Stem Cell Department, AlKhaleej Clinics. Collection of data will be started after the scientific and ethical approval from Dow University, Karachi. After screening by physician and fulfilling the inclusion and exclusion criteria, patients (n=48) will be enrolled. After briefing about the objectives and obtaining formal consent, data will be collected. Participants will be randomized and equally distributed into two groups i.e., twenty-four in control group '1' and twenty-four in treatment group '2'. The control group '1' will receive forward walking in home program after mesenchymal stem cell treatment while the treatment group '2' will be receiving quadriceps isometric exercise, straight limb raises (SLR), hip isometric adductor, knee terminal extension, semi wall squat, quadriceps drill exercises for knee osteoarthritis after mesenchymal stem cell therapy. Treatment plan will be of 8 weeks with 3 sessions in one week for 30 minutes. A physical therapist will do the assessment at baseline and at the end of treatment, other than the principal investigator to measure outcomes by using KOOS score, manual muscle testing and VAS scale. For the completion of the study 6 months are required after synopsis approval.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of age 40 years and above.
* Male and female both will be included.
* Patients with single or both knee OA.
* Patients who had mesenchymal stem cell transplantation.
* Kellgren and Lawrence grade II, III on radiological findings.

Exclusion Criteria:

* Patients with any neurological disorder.
* Any musculoskeletal deformity (varus/valgus).
* Patients who have had any type of lower limb internal fixation.
* Patients who have had any type of lower limb arthroplasty or other knee surgery in the past.
* Patients with a history of any infectious or malignant condition.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-11-06 (Estimated); Study Completion 2023-12-06 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (change is being assessed) | Baseline and 8 weeks
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a self reported specific joint measure developed to assess a broad spectrum of patients with knee injuries and OA, for pain and other symptoms, function in daily life, function in sports and recreation, and quality of knee-related life, being easy to use, evaluating the short- and long-term health problems related to the knee joint.
  The Knee injury and Osteoarthritis Outcome Score contains 42 items covering five subscales: pain, other symptoms, activities of daily living, sports/recreation, and quality of life. A patient's maximum score is 100, which indicates that they have no knee concerns. The lowest possible score is 0, which indicates serious knee issues.

SECONDARY OUTCOMES:
Visual analog scale (change is being assessed) | Baseline and 8 weeks
  It measures the subjective of pain ranges from 10-cm lines with defined cut off scores. The correlation between vertical and horizontal orientations of the VAS is 0.99 . Aggregate score ranges for this screening tool starting with 0-10. Scores between 0-4 means mild pain. Scores between 4-7 indicates moderate pain. Scores between 7-10 means severe pain. pain severity will be assessed at rest and during stairs ascending and descending
Manual Muscle Testing (change is being assessed) | Baseline and 8 weeks
  It is used to assess weakness and is capable of distinguishing actual weakness from imbalance or insufficient endurance. Muscle strength testing is used to assess a complaint of weakness, which commonly occurs when a suspected neurologic condition or muscle weakness is present. The Oxford Scale is the most widely used way of determining muscle strength (AKA Medical Research Council Manual Muscle Testing scale). This method entails putting important muscles in the upper and lower limbs to the test against the examiner's resistance and assessing the patient's strength on a scale of 0 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Farhan I Khan, PhD, Study Director — Dow University of Health Sciences
Locations (2):
- Pakistan (2):
  - Dow Institute of Physical Medicine and Rehabilitation, DUHS., Karachi, Sindh
  - Alkhaleej Ortho Stem Cell Clinic, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No